CLINICAL TRIAL: NCT04508257
Title: Randomized, Double-blind, Parallel, Controlled Study to Evaluate the Nutritive Effects of Two Staged Infant Formulas on Growth and Cognitive Outcomes in Healthy Term Infants
Brief Title: The Effect of a New Infant Formula on Growth and Cognition in Healthy Term Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19-SM-09-FEIHE-001
Record Dates: First submitted 2020-08-02; First posted 2020-08-11 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Child Development
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational Formula (Stage 1&2) (Experimental): Investigational formula contains DHA，ARA and enriched whey protein (source of milk fat globule membrane) to support the healthy growth and Cognitive development of infants.
  Interventions: Dietary Supplement: Oral feeding of Investigational Formula (Stage 1&2)
- Control formula (Stage 1&2) (Active Comparator): Control formula have comparable macronutrients and micronutrients, but does not contain DHA，ARA and MFGM.
  Interventions: Dietary Supplement: Oral feeding of Control formula (Stage 1&2)
- Breast feeding (Other): Breast fed of human milk
  Interventions: Dietary Supplement: Breast feeding

INTERVENTIONS:
Dietary Supplement: Oral feeding of Investigational Formula (Stage 1&2) — Participants will receive stage 1 formulas up to 180 days of age and then switch to stage 2 formulas though 365 days of age.
  Arms: Investigational Formula (Stage 1&2)
Dietary Supplement: Oral feeding of Control formula (Stage 1&2) — Participants will receive stage 1 formulas up to 180 days of age and then switch to stage 2 formulas though 365 days of age.
  Arms: Control formula (Stage 1&2)
Dietary Supplement: Breast feeding — Exclusively breastfed for the first 4 months and continue with supplement food without any marketed infant formula.
  Arms: Breast feeding

SUMMARY:
This study is a multicenter, double-blind, randomized, controlled, parallel-designed, prospective trial and is intended to evaluate the nutritive effects of two staged study formulas on growth and cognitive outcomes. Approximately 450 participants will be enrolled with the expectation of having 105 participants per group (315 for three groups: control group, investigational group, and breastfeeding reference group ) complete Study Visit 6 at 365 days of age ± 7 days (allowing for a 30% drop-out rate). Participants will receive stage 1 formulas up to 180 days of age and then switch to stage 2 formulas though 365 days of age. The study period will include feeding up to 365 days of age and cognitive testing up to 365 days of age. Stool samples will be collected from a subset of participants at enrollment and at 120 days of age for fecal microbiome analysis.

DETAILED DESCRIPTION:
Primary Objective

* Compare measures of normal, healthy mental development at 365 days of age among infants receiving an investigational formula, infants receiving the control and breastfed group.

Secondary Objectives

To compare between the two study groups:

* Measures of mental development up to 365 days of age
* Rate of body weight, length and head circumference gain
* Achieved weight, length and head circumference
* Stool characteristics, tolerance and formula acceptance
* Fecal microbiome analysis
* Antibiotic treatment
* Medically-confirmed adverse

ELIGIBILITY:
Inclusion Criteria:

* 30 days of age at randomization, inclusive (day of birth is considered day 0)
* Exclusively formula-fed for at least 3 days prior to randomization
* Singleton birth
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age)
* Birth weight of 2500g to 4000g
* Signed informed consent obtained for infant's participation in the study
* Parent or guardian of infant agrees not to enroll infant in another interventional clinical research study while participating in this study

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
* Weight at Visit 1 is <95% of birth weight [(weight at Visit 1÷birth weight) x 100 <95%]
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury such as Microcephaly, Macrocephaly or others.
* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
* Weight at Visit 1 is <95% of birth weight [(weight at Visit 1÷birth weight) x 100 <95%]
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury such as Microcephaly, Macrocephaly or others.

Additional Criteria for Inclusion in the Stool Collection Subset

* Vaginal birth
* Participant has not received antibiotic treatment antibiotic and/or corticosteroid treatment for at least 30 days prior to the collection.
* Participant has not consumed prebiotics/probiotics supplements
* Parent/caregiver has access to a home freezer for sample storage

Ages: 30 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Infant cognitive development | at 365 days of age
  Cognitive Scale of the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used to evaluate infant cognitive development at 365 days of age.
  1. Unabbreviated scale title： Bayley-III Scales of Infant Development Tables and Graphs Report-- Cognitive Scale ；
  2. Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  3. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Infant Language capabilities | at 365 days of age
  Language Scale of Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used to evaluate the infant Language capabilities at 365 days of age.
  1. Unabbreviated scale title：Bayley-III Scales of Infant Development Tables and Graphs Report-- Language Scale ；
  2. Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  3. Higher scores mean a better outcome.
Infant motor skills | at 365 days of age
  Motor Scale of Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used to evaluate the infant motor skills at 365 days of age.
  1. Unabbreviated scale title：Bayley-III Scales of Infant Development Tables and Graphs Report-- Motor Scale
  2. Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  3. Higher scores mean a better outcome.
Infant social-emotional capabilities | at 365 days of age
  Social-emotional Scale of Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used to evaluate the infant social-emotional capabilities at 365 days of age.
  1. Unabbreviated scale title：Bayley-III Scales of Infant Development Tables and Graphs Report-- Social-emotional Scale.
  2. Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  3. Higher scores mean a better outcome.
Infant adaptive behavior tests | at 365 days of age
  Adaptive behavior Scale of Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used as the infant adaptive behavior assessment tool at 365 days of age.
  1. Unabbreviated scale title：Bayley-III Scales of Infant Development Tables and Graphs Report-- Adaptive behavior scale
  2. Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  3. Higher scores mean a better outcome.
Ages and Stages Questionnaires (ASQ) | at 120, 180, and 275 days of age
  Ages and Stages Questionnaires (ASQ) is administered at 120, 180, and 275 days of age.
  ASQ is a developmental screening system comprised of age-specific questionnaires which measure 5 domains of infant development.
  1. Unabbreviated scale title： Ages and Stages Questionnaires；
  2. the minimum~maximum value：0~60 points；
  3. Higher scores mean a better outcome.
MacArthur-Bates Communicative Development Inventory（CDI） tests | at 365 days of age
  MacArthur-Bates Communicative Development Inventory (CDI) tests is administered at 365 days of age.
  It is a parent-report measure that has been validated against actual child language diaries.
  1. Unabbreviated scale title：MacArthur-Bates Communicative Development Inventory evaluation form
  2. the minimum~maximum percentile：5%-99%；
  3. The higher the percentile, the better；
Carey Toddler Temperament Scale( TTS )tests | at 365 days of age
  Carey Toddler Temperament Scale (TTS) tests is administered at 365 days of age. TTS is a 97-item questionnaire which measures the nine categories of temperament: activity level, regularity, adaptability, approach-withdrawal, intensity, mood, persistence, sensory threshold and distractibility.
  1. Unabbreviated scale title：Carey Toddler Temperament Scale
  2. Normal score range of TTS for 1 to 3 year old infants:
     Activity: 12.4 ~ 19.6 Fitness: 6.5 ~ 11.9 Emotional nature: 8.9 ~ 14.1 Regularity: 8 ~ 13 intensity: 11.5 ~ 18.1 Degree of distraction: 8 ~ 12.4 Below or above the normal range are temperament bias.
  3. Temperament is innate and there is no difference between good and bad. infants with different temperament need different care.
Infant attention | at 365 days of age
  Single object attention and free play tasks is used to measure the infant's attention capabilities. The tasks assess overall fixation (attention) and looking away (inattention) in regards to novel and familiar objects.
Achieve body weight | at 30, 90, 120, 180, 275, and 365 days of age
  Achieve body weight (grams) of infants and toddlers at each study visit
Achieve body length | at 30, 90, 120, 180, 275, and 365 days of age
  Achieve body length (cm) of infants and toddlers at each study visit
Achieve head circumference | at 30, 90, 120, 180, 275, and 365 days of age
  Achieve head circumference (cm) of infants and toddlers at each study visit
24-Hour dietary recall of Formula intake | at 30, 90, 120, 180, 275, and 365 days of age
  The parent/caregiver need to record the amount of study formula consumed as well as any other infant formula or milk consumed since the last study visit
24-Hour Recall of Stool Characteristics Questionnaire | at 30, 90, 120, 180, 275, and 365 days of age
  The parent/caregiver will also be asked to recall the number of bowel movements and the stool consistency seen most often over the 24-hour period. Pictures will be provided to the participant's parent or caregiver for use as a guide in rating the stool consistency.
  Questionnaire: What stool consistency was seen most often in your baby's bowel movements over the past 24 hours?(Use pictures provided for reference) (0) No bowel movement;
  1. Hard- dry, hard pellets;
  2. Formed- definite shape, not dry;
  3. Soft-no definite shape, pasty;
  4. Unformed or seedy- no shape, some water or small lumps ;
  5. Waterly- no shape, mainly water
  For option 0~5, 0 and 1 represent poor stool Characteristics , 2-5 represent fine stool Characteristics.
24-Hour Recall of Tolerance Questionnaire | at 30, 90, 120, 180, 275, and 365 days of age
  Tolerance information concerning how fussy and gassy the infant has been and if the infant has been more fussy and/or gassy than normal need to be recalled and recorded by parent/caregiver for the 24-hour period prior to the study visit.
  Questionnaire:
  1. Over the past 24 hours, how fussy has your baby been? (0) Not at all fussy; (1)Slightly fussy; (2) Moderately fussy; (3) Very fussy; (4) Extremely fussy;
  2. Over the past 24 hours, ____ was your baby? (0) Less fussy than normal ; (1) About the same level of fussiness as always; (2) More fussy than normal
  3. Over the past 24 hours, how much gas has your baby had? (0) Not at all ; (1) Slightly amount of gas; (2) Moderate amount of gas; (3) Excessive amount of gas
  4. Over the past 24 hours, did your baby have : (0) Less gas than normal; (1) About the same amount of gas as normal ; (2) More gas than normal
  For Question 1 ~ 4, the lower the score, the better.
Percentages of adverse events | from 30 days of age to 365 days of age
  Number and percentages of infants in each group experiencing any medically-confirmed adverse events and any serious adverse events.
  1. A medically-confirmed adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding that is considered clinically relevant by the Health Care Provider), including eyes, ear, nose and throat and the whole body manifestations, respiratory manifestations, dermatologic manifestations, Musculoskeletal manifestations, Metabolism and nutrition manifestations,etc.
  2. An adverse event is considered serious if it meets one or more of the following criteria:
     * results in death
     * is life-threatening
     * requires inpatient hospitalization or prolongation of existing hospitalization
     * results in persistent or significant disability/incapacity, or
     * is a congenital anomaly/birth defect
Stool collection | at enrollment and 120 days of age
  Fecal microbiome analysis of samples collected at enrollment and at 120 days of age
Percentage of infants with oral antibiotic treatments | at 365 days of age
  Percentage(%) of infants in each group using any oral antibiotic treatments.
Percentage of infants with intramuscular antibiotic treatments | at 365 days of age
  Percentage(%) of infants in each group using intramuscular antibiotic treatments.
Percentage of infants with intravenous (IV) antibiotic treatments | at 365 days of age
  Percentage(%) of infants in each group using intravenous (IV) antibiotic treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Zhang, M.D., Ph.D., Principal Investigator — Anhui Medical University Affiliated Children's Hospital, China
Locations (3):
- China (3):
  - Jinhua Nanyuan Community Health Center (site 1919), Jinhua, Zhejiang
  - Jinhua Qiubin Community Health Center (site 1969), Jinhua, Zhejiang
  - Jinhua Xiguan Community Health Center (site 1966), Jinhua, Zhejiang